CLINICAL TRIAL: NCT05200832
Title: Impact of Long COVID-19 on the Health and Quality of Life of Military Personnel (Active or Retired) and Their Families
Acronym: IMP@LA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2021PPRC06; 2021-A02623-38 (Other: IDRCB)
Record Dates: First submitted 2022-01-19; First posted 2022-01-21 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: COVID-19
Keywords: quality of life; long COVID
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID+: Participants who have experienced COVID-19
  Interventions: Other: Online questionnaire; Other: Semi-structured interview
- COVID-: Participants who have not experienced COVID-19
  Interventions: Other: Online questionnaire; Other: Semi-structured interview

INTERVENTIONS:
Other: Online questionnaire — Participants will be asked to complete an online questionnaire about their health and quality of life since the start of the pandemic.
Other: Semi-structured interview — 20 participants (10 from each group) will be randomly selected to participate in a semi-structured interview focusing on their perception of their health and quality of life since the start of the pandemic.

SUMMARY:
Severe and sometimes irreversible sequelae are observed in people who have developed a severe form of COVID-19 (pulmonary, cardiovascular, renal, neurological sequelae among others). More than 10% of individuals who contracted the disease, even in a mild form, still have at least one of the initial symptoms at six months, also known as prolonged symptoms or long COVID syndrome. The most frequently observed symptoms are asthenia, neurological disorders (headache, anosmia, ageusia, etc.), cardio-thoracic disorders, pain, digestive or skin disorders. Very recently, the first results of a British prospective cohort study (PHOSPCovid) indicate that more than half of the COVID-19 survivors who were hospitalised experienced a very severe to moderate deterioration in their mental and/or physical health five months after hospitalisation. Women are particularly affected. Another American study shows that 85% of non-hospitalised COVID-19 patients developed at least 4 neurological symptoms impacting their quality of life. The most common are: "brain fog" (81%), headaches (68%), numbness or tingling (60%), taste impairment (59%) and loss of smell (55%).

These disabling symptoms may persist for weeks or months, deteriorating the quality of life of patients and making it difficult for some to return to a normal life. On the basis of current knowledge concerning the long-term sequelae of SARS-CoV-2 infection, it seems necessary to offer these subjects a specific care pathway and to adapt their living and working conditions beyond their medical care.

The present study is aimed at measuring the impact of long COVID on the health and quality of life of the defence community (military personnel and their families).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years-old
* Be affiliated to the French military health insurance

Exclusion Criteria:

* Age < 18 years-old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of people affiliated to the French military health insurance, i.e., military Personnel (active or retired) and their families.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-09-05 (Estimated); Study Completion 2023-09-05 (Estimated)

PRIMARY OUTCOMES:
Prevalence of mental health events | Until the end of the study (12 months)
  Prevalence of mental health events will be calculated in each group, the compared:
  number of participants who report having experienced a mental health event (e.g. anxiety disorder) divided by the number of participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Epidémiologie et de Santé Publique des Armées, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided